CLINICAL TRIAL: NCT03536013
Title: A Clinical Investigation Evaluating Efficacy of a Full-Thickness Placental Allograft in Lumbar Microdiscectomy Outcomes
Brief Title: Efficacy of a Full-Thickness Placental Allograft in Lumbar Microdiscectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: StimLabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSP17-002
Record Dates: First submitted 2018-04-30; First posted 2018-05-24 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Surgical Wound; Herniation
MeSH Terms: conditions — Surgical Wound; Hernia

STUDY DESIGN:
Intervention Model Description: Blind study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 91 patients will undergo a typical lumbar microdiscectomy with the addition of a full-thickness placental allograft after the microdiscectomy has been performed.
  Interventions: Other: Other: Full-thickness placental allograft
- Control (No Intervention): 91 patients will undergo a typical lumbar microdiscectomy without the addition of a full-thickness placental allograft.

INTERVENTIONS:
Other: Other: Full-thickness placental allograft — A full-thickness placental allograft will be applied to the annulus of the index lumbar level prior to site closure.
  Arms: Treatment

SUMMARY:
To evaluate the efficacy of full thickness placental allograft use in Microdiscectomy application. To evaluate post-microdiscectomy reherniation rate in patients treated with full-thickness placental allografts.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of full thickness placental allograft use in improving back and leg pain, when applied to patients undergoing lumbar microdiscectomy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory with radiating low back and leg pain for greater than 6 months prior to surgery with clinical diagnosis of lumbar protruding disc.
* Consent and compliance with all aspects of the study protocol, methods, providing data during follow-up contact.

Exclusion Criteria:

* Severe hypertension systolic blood pressure (greater than or equal to 200 mm -Hg or diastolic blood pressure greater than or equal to 182 mm Hg)
* BMI greater than 45 kg/m2
* Subject has had major surgery at the index level
* Is an active smoker or stopped smoking in the last 6 months
* Any pain that could interfere with the assessment of index level pain (e.g. pain in any other part of the spine)
* Active rheumatoid arthritis
* Active, local or systemic malignancy such as lung cancer or leukemia
* History of vascular disease or sickle cell anemia
* Use of the following medications:

No significant anticoagulant therapy (e.g. Heparin or Lovenox) during the study (treatment such as Aspirin and Plavix are allowed)

* No systemic treatments that may interfere with safety or efficacy assessments during the study
* No immunosuppressants
* No use of corticosteroids

  * Subject is pregnant or plans to become pregnant within 24 months of treatment
  * Subject does not provide full consent
  * Personal injury, workman's compensation or other legally-related treatment patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Measuring efficacy of full-thickness placental allograft in reducing back and leg pain post-microdiscectomy. | 24 months
  Oswestry Disability Index (ODI)
Measuring efficacy of full-thickness placental allograft in reducing back and leg pain post-microdiscectomy. | 24 months
  12-Item Short Form Survey (SF12)

SECONDARY OUTCOMES:
Evaluation of post-microdiscectomy reherniation rate. | 24 month
  Reherniation rates will be compared between the experimental and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Morrison, M.D., Principal Investigator — Polaris Spine and Neurosurgery
Locations (1):
- Polaris Spine and Neurosurgery, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The sponsor will not have access to personally identifying participant information.